CLINICAL TRIAL: NCT00000839
Title: A Phase I Trial to Evaluate Didanosine (ddI) in HIV-Infected Pregnant Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 249; 11226 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; Pregnancy
Keywords: Pregnancy Trimester, Third; Pregnancy; Pregnancy Complications, Infectious; Didanosine; Acquired Immunodeficiency Syndrome; AIDS-Related Complex
MeSH Terms: conditions — HIV Infections; Pregnancy Complications, Infectious; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Didanosine

INTERVENTIONS:
Drug: Didanosine

SUMMARY:
To assess the pharmacokinetics, safety, and toxicity of intravenous and oral didanosine (ddI) administration in third trimester pregnant women who are HIV positive but are either intolerant or resistant to zidovudine (AZT). To collect data on infant toxicity following maternal treatment with ddI during the third trimester of pregnancy.

AZT may not be the optimal antiretroviral agent for all pregnant women requiring therapy for HIV infection. Although ddI has been approved for use in HIV-infected adults and older children, the safety and pharmacokinetics of ddI in pregnant women has not yet been determined.

DETAILED DESCRIPTION:
AZT may not be the optimal antiretroviral agent for all pregnant women requiring therapy for HIV infection. Although ddI has been approved for use in HIV-infected adults and older children, the safety and pharmacokinetics of ddI in pregnant women has not yet been determined.

Patients receive a single IV dose of ddI on day 1 and pharmacokinetics values are determined. At least 48 hours but no more than 1 week after the IV dose, patients receive an oral dose, and oral pharmacokinetics are obtained for 8 hours. Oral ddI is then administered every 12 hours until labor commences and then after delivery, every 12 hours until 6 weeks postpartum. During labor and delivery, patients receive a loading dose of ddI followed by continuous infusion. Pharmacokinetics are obtained during infusion and also at 6 weeks postpartum. AS PER AMENDMENT 11/24/97: Maternal IV pharmacokinetic studies will not be performed after ddI IV formulation has expired (11/30/97). Maternal and cord samples will be required regardless of whether mother has received continuous IV ddI during labor.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Aerosolized pentamidine.
* IV AZT during labor.

Patients must have:

* HIV infection.
* CD4 count > 50 and < 350 cells/mm3.
* AZT intolerance or resistance.
* Gestational age at least 26 weeks but not more than 36 weeks.
* Consent of guardian if necessary. The father of the fetus must also provide consent if available after reasonable attempts have been made to contact him.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Multiple gestation.
* Current obstetrical complication, such as major anomalies, growth retardation, abnormal fluid level, fetal hydrops, or placental abruption (placenta previa is allowed).
* No access to a participating ACTU.

Concurrent Medication:

Excluded:

* Drugs that might aggravate pancreatitis, such as steroids, isoniazid, and parenteral pentamidine.
* Antiretrovirals other than ddI (although IV AZT is allowed during labor).

Patients with the following prior conditions are excluded:

* History of stillbirth, neonatal loss, or previous infant with anomaly (history of preeclampsia or preterm labor is permitted).
* History of maternal medical complications including but not limited to malabsorption syndrome, pancreatitis, neurological complications including grade 2 or worse peripheral neuropathy, symptomatic cholelithiasis, or prior active CMV disease requiring ganciclovir or foscarnet.
* History of poor medical compliance not related to access to medical care.

Prior Medication:

Excluded:

* ddI within 24 hours prior to study entry.

Min Age: 13 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12
Dates: Study Completion 2001-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Livingston E, Study Chair; Bartlett JA, Study Chair; Unadkat J, Study Chair
Locations (13):
- United States (11):
  - UCLA-Los Angeles/Brazil AIDS Consortium (LABAC) CRS, Los Angeles, California
  - UCSD Maternal, Child, and Adolescent HIV CRS, San Diego, California
  - Univ. of Florida Jacksonville NICHD CRS, Jacksonville, Florida
  - Univ. of Miami Ped. Perinatal HIV/AIDS CRS, Miami, Florida
  - Rush Univ. Med. Ctr. ACTG CRS, Chicago, Illinois
  - Tulane Univ. Health Science Ctr., Tulane Univ. Hosp. & Clinic, New Orleans, Louisiana
  - Tulane/LSU Maternal/Child CRS, New Orleans, Louisiana
  - NJ Med. School CRS, Newark, New Jersey
  - Columbia IMPAACT CRS, New York, New York
  - Incarnation Children's Ctr., New York, New York
  - DUMC Ped. CRS, Durham, North Carolina
- Puerto Rico (2):
  - San Juan City Hosp. PR NICHD CRS, San Juan
  - Univ. of Puerto Rico Ped. HIV/AIDS Research Program CRS, San Juan

REFERENCES:
- [Background] Livingston E, Patil S, Unadkat J, McKinney R, Abreu E, Bardequez A, O'Sullivan M. Placental transfer of didanosine (ddI) and initial evaluation of didanosine toxicity in HIV-1 infected pregnant women and their offspring. Conf Retroviruses Opportunistic Infect. 1998 Feb 1-5;5th:121 (abstract no 226)
- [Background] McKinney RE Jr. Ongoing and future trials of antiretroviral therapy in the pediatric AIDS clinical trials group (PACTG). Conf Retroviruses Opportunistic Infect. 1996 Jan 28-Feb 1;3rd:173
- [Background] Patil SD, Livingston E, McKinney RE, Abreu E, O'Sullivan MJ, Bardequez A, Unadkat JD. Does pregnancy affect the pharmacokinetics of didanosine (ddI) in HIV-1 infected women? Conf Retroviruses Opportunistic Infect. 1998 Feb 1-5;5th:121 (abstract no 225)